CLINICAL TRIAL: NCT02033330
Title: Assessment of Bioavailability of Phenolics From an Orange Peel Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Cordiart-PKA-1
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Improving Bioavailability
Keywords: phenolics; orange peel; bioavailability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- phenolics form orange peel, type 1 (Active Comparator): 1 dose of 500 mg of phenolics from orange peel, orally ingested
  Interventions: Dietary Supplement: phenolics form orange peel
- phenolics from orange peel, type 2 (Active Comparator): 1 dose of 500 mg of phenolics from orange peel, orally ingested
  Interventions: Dietary Supplement: phenolics form orange peel
- phenolics from orange peel, type 3 (Experimental): 1 dose of 500 mg of phenolics from orange peel, orally ingested
  Interventions: Dietary Supplement: phenolics form orange peel

INTERVENTIONS:
Dietary Supplement: phenolics form orange peel

SUMMARY:
In this study, the bioavailability of a specific orange peel extract is tested. The composition and morphology of the test product is altered compared to the generic product, which is used as a control. Due to intellectual property issues, more information cannot be given at this moment. Also the difference in bioavailability between a capsule and a lozenge is tested. The hypothesis is that the bioavailability of the altered extract will be improved compared to the control.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* BMI 18.5 to 25

Exclusion Criteria:

* pregnancy
* smoking
* alcohol or drug abuse
* use of medication
* use of nutritional supplements
* abnormal liver or kidney function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
plasma concentrations of specific phenolics and their metabolites | up to 24 hours

SECONDARY OUTCOMES:
urine concentrations of specific phenolics and their metabolites | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Chris Van der Grinten, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands